CLINICAL TRIAL: NCT02302677
Title: The Effect of Sleeve Gastrectomy on Post-prandial Serum Bile Acids
Acronym: BAS
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0695-14-FB
Record Dates: First submitted 2014-11-19; First posted 2014-11-27 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Obesity
Keywords: bile acids; sleeve gastrectomy; obesity; GLP-1; FGF-19
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective study of meal-induced bile acid physiology before and after sleeve gastrectomy (SG) surgery. Weight loss and metabolic improvement associated with weight loss surgery cannot be entirely attributed to restriction in stomach size and food intake. Bile acids (BAs), amphipathic steroids that have a role in lipid uptake and metabolism in the gastrointestinal tract, are involved in post-prandial glucose homeostasis and energy expenditure & are a potential intermediary in weight loss following bariatric surgery. It is unknown if SG increases post-prandial BAs in humans and if an increase in BA signaling impacts weight loss and co-morbidity resolution after surgery. The investigators hypothesis is that SG will increase the post-prandial serum and urine BAs and that the change in the BA profile is a mechanism for restriction-independent weight-loss following SG. SG patients will undergo a meal challenge pre-operatively, and at 1, 3, and 12 months post-operatively, with measurement of post-prandial serum and urine BAs and downstream hormones, glucagon-like peptide 1 (GLP-1) and fibroblast growth factor 19 (FGF19), and a scoring of satiety before and after the meal challenge using a Visual Analog Scale. Serum insulin, glucose, and C4 levels will also be measured to assess metabolic changes associated with SG. Serum and urine BA levels will be compared to post-operative excess weight loss at 12 months. Before and after each meal challenge, patients will be asked to score satiety, and this will be correlated to weight loss, bile acids, GLP-1, and FGF19.

DETAILED DESCRIPTION:
SUMMARY Bariatric surgeries, such as sleeve gastrectomy (SG), have become an important therapeutic option for morbid obesity and the treatment of obesity-associated co-morbidities.

There is evidence that the weight loss and metabolic improvements associated with SG cannot be entirely attributed to a restriction in stomach size nor nutrient malabsorption. Bile acids (BAs) are a novel potential intermediary in restriction-independent weight loss following SG. Bile acids are amphipathic steroids that have a role in lipid uptake and metabolism in the gastrointestinal tract as well as post-prandial glucose homeostasis and energy expenditure. BAs are the natural ligand for the nuclear farnesoid X receptor (FXR) and the BA activated, cell surface G-protein coupled receptor, TGR5. FXR activation inhibits lipogenesis, glycolysis, BA synthesis and stimulates FGF19 production, which functions in the regulation of BA synthesis. TGR5 activation increases energy expenditure and stimulates the enteroendocrine L cells to secrete the incretin hormone, glucagon-like peptide 1 (GLP-1). Both roux-en-y gastric bypass (RYGB) and SG, unlike gastric banding and dieting, have been shown to paradoxically increase energy expenditure and augment post-prandial GLP-1 secretion, suggesting a restriction-independent mechanism of weight-loss possibly mediated by changes in BA signaling [1-4]. Although suggested by animal models of SG, it is currently unknown if SG increases post-prandial BAs in humans and if an increase in BA signaling impacts weight loss and co-morbidity resolution following surgery. The identification of restriction-independent mechanisms of weight loss after SG may lead to the development of novel surgical or medical therapies that exploit these specific mechanisms to achieve significant and sustainable weight loss in morbidly obese patients. Further, understanding the mechanisms of weight loss after SG may lead to the identification of patients pre-operatively or early in the post-operative period who are at high risk for poor surgical weight loss outcomes. The proposed work is a prospective study of meal-induced BA physiology before and after SG.

The investigators hypothesize that SG will increase the post-prandial serum and urine BAs and that the change in the post-operative bile acid profile is a mechanism for restriction independent weight-loss following sleeve gastrectomy.

The investigators first specific aim is to determine the effect of SG on post-prandial total BAs and BA subtypes. The investigators working hypothesis is that SG will increase post-prandial total BAs as well as modulate specific BA subtypes. Eligible SG patients will undergo a meal challenge preoperatively, and at one, three, and 12 months post-operatively, with measurement of postprandial serum and urine bile acids by ultra-performance liquid chromatography and mass spectroscopy (UPLC/MS) as well as GLP-1 and FGF19 by ELISA. Serum insulin, glucose, and C4 levels will also be measured to assess metabolic changes associated with SG.

The investigators second specific aim is to correlate the changes in post-prandial bile acids and bile acid subtypes after SG to post-operative excess weight loss and satiety. The investigators working hypothesis is that post-prandial BAs and BA subtypes will increase following SG, and the increase in bile acids will correspond to post-operative excess weight loss, GLP-1 production, and meal satiety. Post-prandial serum and urine BAs preoperatively and at 1, 3, and 12 months following SG will be compared to post-operative excess weight loss at 12 months. Before and after each meal challenge, patients will be asked to score satiety, and these scores will be correlated to excess weight loss, GLP-1 and total BA as well as BA subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years of age and ≤ 70 at the time of surgery
2. Participant in the Surgical Weight Loss Program of the Bariatrics Center of UNMC
3. SG approved to be completed at UNMC
4. Primary bariatric surgery or prior band placement and removal over 2 years prior

Exclusion criteria:

1. Past medical history of small bowel resection or right colectomy
2. History of cirrhosis
3. Current or planned use of bile acid sequestrants
4. Bariatric surgery being performed as a revisional procedure other than #4 as above. -

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients who are being treated in the Bariatric Clinic at the University of Nebraska Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Measurement of serum bile acids and correlation to weight loss and satiety. | 1 year
  Serum bile acids will be measured prior to surgery and at 1, 3 and 12 months post-surgery. The level of this compound will be compared to weight loss and satiety.
Measurement of urine bile acids and correlation to weight loss and satiety. | 1 year
  Urine bile acids will be measured prior to surgery and at 1, 3 and 12 months post-surgery. The level of this compound will be compared to weight loss and satiety.
Measurement of serum GLP-1 and correlation to weight loss and satiety. | 1 year
  Serum GLP-1 will be measured prior to surgery and at 1, 3 and 12 months post-surgery. The level of this compound will be compared to weight loss and satiety.
Measurement of serum FGF-19 and correlation to weight loss and satiety. | 1 year
  Serum FGF-19 will be measured prior to surgery and at 1, 3 and 12 months post-surgery. The level of this compound will be compared to weight loss and satiety.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Kindel, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No